CLINICAL TRIAL: NCT02895217
Title: Evaluation of Energy Balance During Aquatic Cycling Exercise in Premenopausal Women: Effect of Body Composition Status
Brief Title: Aquatic Exercise and Metabolism in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0272; 2016-A00197-44 (Other: 2016-A00197-44)
Record Dates: First submitted 2016-07-12; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Aquacycling
Keywords: Energy expenditure; Food intake; Women; aquacycling

ARMS (2):
- Cycling exercise in water (Experimental): The aim of this project is to investigate energetic response (energy expenditure and food intake) of a single bout of cycling exercise in water vs on dryland in normal weight and overweight premenopausal women.
  Interventions: Other: ergocycle
- cycling exercise on dryland (Experimental): The aim of this project is to investigate energetic response (energy expenditure and food intake) of a single bout of cycling exercise in water vs on dryland in normal weight and overweight premenopausal women.
  Interventions: Other: ergocycle

INTERVENTIONS:
Other: ergocycle

SUMMARY:
Exercise training on an immersible ergocycle is becoming more popular as it appears to be more suitable for men and women even with poor physical activity level. Commercial tagline highlight beneficial effect of this activity on weight management. However there are poor information concerning the energy response induced by this activity. The aim of this project is to investigate energetic response (energy expenditure and food intake) of a single bout of cycling exercise in water vs on dryland in normal weight and overweight premenopausal women.

DETAILED DESCRIPTION:
After inclusion visit, all subject will be submitted to DXA to obtain body composition data. Then subjects will be submitted to four experimental session in a semi-randomized order. For all those session, subjects will take a standardized breakfast (570kcal) three hours before experimental session.

Control session (CON): subject will stand sited without any activity during 30 min.

Water exercise session (WAT): subject will exercise on an immersed ergocycle during 30 min at 50 rpm.

Dryland session 1 (LAND-1): subject will exercise on dryland, on the same ergocycle than in WAT session, during 30 min at 50 rpm.

Dryland session 2 (LAND-2): subject will exercise on dryland on the same ergocycle than in WAT. Intensity of exercise will be set at the same heart rate average than in WAT session, exercise will be stopped when subject will have reached the same energy expenditure than during WAT session.

During each session, energy expenditure, heart rate and rate of perceived exertion will be measured at 15 min and 30min.

Appetite and hunger sensation will be measured with a specific scale at different time point of each day of experimental session. Thirty minutes after the end of each experimental session subjects will have a buffet meal for lunch time.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 23 and 40 years
* BMI under 25kg.m2 for normal weight women and between 25 and 29,9 kg.m2 for overweight women
* Daily breakfast
* Subject which approved informed consent
* Subject with French medical affiliation

Exclusion Criteria:

* Specific medical treatment
* Aquaphobia
* Subject under specific diet regimen or weight loss program
* Subject with cardio-vascular disease
* Surgical intervention less than 3 months
* Subject refusing informed and written consent
* Subject without French medical affiliation
* subject refusing inscription to the national voluntary list
* subject being in an exclusion period
* subject smoking or drinking alcohol frequently
* subject with intense physical activity

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Food intake during buffet meal | at day 1
  during buffet meal 30 min after the end of each experimental session

SECONDARY OUTCOMES:
Appetite sensation | at day 1
  during each session (before and after breakfast, before and after experimental session, 30 min after the experimental session, 30min after the end of buffet meal at lunch time) . Each sensation is measured with a visual analogue scale
Energy expenditure in kcal | at day 1
  during each session (during each 30min session measured by indirect calorimetry)
Rate of perceived exertion | at day 1
  during each session
hunger sensation | at day 1
  during each session( before and after breakfast, before and after experimental session, 30 min after the experimental session, 30min after the end of buffet meal at lunch time)

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Brechat PH, Wolf JP, Simon-Rigaud ML, Brechat N, Kantelip JP, Berthelay S, Regnard J. Influence of immersion on respiratory requirements during 30-min cycling exercise. Eur Respir J. 1999 Apr;13(4):860-6. doi: 10.1034/j.1399-3003.1999.13d28.x. PMID 10362054